CLINICAL TRIAL: NCT01174446
Title: Recombinant Factor IX (BAX 326): A Phase 1/3, Prospective, Controlled, Multicenter Study Evaluating Pharmacokinetics, Efficacy, Safety and Immunogenicity in Previously Treated Patients With Severe or Moderately Severe Hemophilia B
Brief Title: Pivotal Study (Pharmacokinetics, Efficacy, Safety) of BAX 326 (rFIX) in Hemophilia B Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 250901; 2009-016720-31 (EudraCT Number)
Record Dates: First submitted 2010-08-02; First posted 2010-08-03 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BAX 326 (Experimental): Recombinant factor IX (rFIX)
  Interventions: Biological: BAX 326
- BeneFIX (Active Comparator): Recombinant Factor IX (rFIX)
  Interventions: Biological: BeneFIX

INTERVENTIONS:
Biological: BAX 326 — * Study Part 1: Pharmacokinetic (PK) Crossover with BAX326 and BeneFIX
  * Study Part 2: Open-label evaluation of prophylaxis and on-demand BAX326 only
  * Study Part 3: Open-label repeat of PK evaluation (repeat Study Part 1) with BAX326 only and same study participants as Study Part 1
  Other Names: Recombinant factor IX (rFIX); RIXUBIS
  Arms: BAX 326
Biological: BeneFIX — * Study Part 1: Pharmacokinetic (PK) Crossover with BAX326 and BeneFIX.
  * BeneFIX only used in Part 1 of this study.
  * Study Part 2 and 3 only utilized BAX326
  Other Names: Recombinant factor IX (rFIX)
  Arms: BeneFIX

SUMMARY:
The purpose of this pivotal Phase 1/3 study is to determine the pharmacokinetic (PK) parameters, the hemostatic efficacy, and the safety of BAX 326, a recombinant factor IX, in previously treated patients (PTPs) with severe and moderately severe hemophilia B.

ELIGIBILITY:
Main Inclusion Criteria:

* Participant is 12 to 65 years old at the time of screening
* Participant and/or legal representative has/have provided signed informed consent
* Participant has severe (factor IX (FIX) level < 1%) or moderately severe (FIX level 1-2%) hemophilia B (based on the one stage activated partial thromboplastin time (aPTT) assay), as tested at screening at the central laboratory
* Participant is previously treated with plasma-derived or recombinant FIX concentrate(s) for a minimum of 150 exposure days (EDs) (based on the participant's medical records); if a verifiable, documented history is unavailable, the participant can be enrolled if s/he has 100-150 EDs to any FIX product that are not fully documented and has participated in Study 050901 for at least 50 EDs to Immunine prior to enrollment (not valid for US and Japan).
* Participant has no evidence of a history of FIX inhibitors
* If the participant is to receive prophylactic treatment, the participant is willing to receive prophylactic treatment over a period of 6 months.
* If the participant is to receive on-demand treatment, the participant has ≥12 documented bleeding episodes requiring treatment within 12 months prior to enrollment and is willing to receive on-demand treatment for the duration of this study.

Main Exclusion Criteria:

* The participant has a history of FIX inhibitors with a titer ≥0.6 Bethesda Units (BU) (as determined by the Nijmegen modification of the Bethesda assay or the assay employed in the respective local laboratory) at any time prior to screening
* The participant has a detectable FIX inhibitor at screening, with a titer ≥0.6 BU as determined by the Nijmegen modification of the Bethesda assay in the central laboratory
* The participant's weight is < 35 kg or > 120 kg
* The participant has a history of allergic reaction, eg, anaphylaxis, following exposure to FIX concentrate(s)
* The participant has a known hypersensitivity to hamster proteins or recombinant furin (rFurin)
* The participant has ongoing or recent evidence of a thrombotic disease, fibrinolysis or disseminated intravascular coagulation (DIC)

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-07-29 (Actual); Primary Completion 2012-05-03 (Actual); Study Completion 2012-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (25):
- Rosario, Argentina
- Brazil (2):
  - Brasília
  - São Paulo
- Sofia, Bulgaria
- Santiago, Chile
- Colombia (2):
  - Bogotá
  - Cali
- Prague, Czechia
- Japan (4):
  - Hiroshima
  - Nara
  - Tochigi
  - Tokyo
- Poland (4):
  - Gdansk
  - Krakow
  - Lodz
  - Warsaw
- Romania (2):
  - Bucharest
  - Timișoara
- Russia (3):
  - Kirov
  - Moscow
  - Saint Petersburg
- Barcelona, Spain
- Malmo, Sweden
- Lviv, Ukraine
- London, United Kingdom

REFERENCES:
- [Result] Windyga J, Lissitchkov T, Stasyshyn O, Mamonov V, Rusen L, Lamas JL, Oh MS, Chapman M, Fritsch S, Pavlova BG, Wong WY, Abbuehl BE. Pharmacokinetics, efficacy and safety of BAX326, a novel recombinant factor IX: a prospective, controlled, multicentre phase I/III study in previously treated patients with severe (FIX level <1%) or moderately severe (FIX level </=2%) haemophilia B. Haemophilia. 2014 Jan;20(1):15-24. doi: 10.1111/hae.12228. Epub 2013 Jul 9. PMID 23834666

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 29 clinical sites in South America, Europe, and Japan.
Pre-assignment Details: 86 enrolled. 1 withdrew consent prior to randomization. -31 were enrolled and randomized in Parts 1-3. Prior to receiving study drug: 3 discontinued by participant. -Part 2 an additional 54 were enrolled. Prior to receiving study drug: 3 discontinued by participant, 1 withdrew due to an AE, 2 screen failures, and 3 withdrew due to site closure.
Groups:
- PK (BAX326 Then BeneFIX) Then Prophylaxis Then PK BAX326 Only: -Study Part 1: Pharmacokinetic (PK) Crossover with BAX326 (75 ± 5 IU/kg) then BeneFIX (75 ± 5 IU/kg). -Study Part 2: Open-label evaluation of prophylaxis and on-demand BAX326 only -Study Part 3: Open-label repeat of PK evaluation (repeat Study Part 1) with BAX326 (75 ± 5 IU/kg) only and same study participants as Study Part 1
- PK (BeneFIX Then BAX326) Then Prophylaxis Then PK BAX326 Only: -Study Part 1: Pharmacokinetic (PK) Crossover with BeneFIX (75 ± 5 IU/kg) then BAX326 (75 ± 5 IU/kg). -Study Part 2: Open-label evaluation of prophylaxis and on-demand BAX326 only -Study Part 3: Open-label repeat of PK evaluation (repeat Study Part 1) with BAX326 (75 ± 5 IU/kg) only and same study participants as Study Part 1
- Study Part 2 Only: BAX326 Prophylaxis; Study Part 2 Only: BAX326 On-Demand: -Participants were only in Study Part 2 (i.e., did not participate in Study Parts 1 and 3)
Period: Part 1 -Pharmacokinetic Crossover
Arm/Group | PK (BAX326 Then BeneFIX) Then Prophylaxis Then PK BAX326 Only | PK (BeneFIX Then BAX326) Then Prophylaxis Then PK BAX326 Only | Study Part 2 Only: BAX326 Prophylaxis | Study Part 2 Only: BAX326 On-Demand
Started | 14 | 14 | 0 | 0
Completed | 14 (BAX326 was mistakenly infused for second PK infusion (ie should have been BeneFIX) for 1 participant) | 14 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2 -BAX326 Prophylaxis and On-demand
Arm/Group | PK (BAX326 Then BeneFIX) Then Prophylaxis Then PK BAX326 Only | PK (BeneFIX Then BAX326) Then Prophylaxis Then PK BAX326 Only | Study Part 2 Only: BAX326 Prophylaxis | Study Part 2 Only: BAX326 On-Demand
Started | 14 (In Study Part 2 all 14 participants received Prophylaxis) | 14 (In Study Part 2 all 14 participants received Prophylaxis) | 31 (This group only participated in Study Part 2) | 14 (This group only participated in Study Part 2)
Completed | 14 | 14 | 29 | 14
Not Completed | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Period: Part 3 -Pharmacokinetic BAX326 Only
Arm/Group | PK (BAX326 Then BeneFIX) Then Prophylaxis Then PK BAX326 Only | PK (BeneFIX Then BAX326) Then Prophylaxis Then PK BAX326 Only | Study Part 2 Only: BAX326 Prophylaxis | Study Part 2 Only: BAX326 On-Demand
Started | 14 (Includes all participants who completed Part 1) | 14 (Includes all participants who completed Part 1) | 0 | 0
Completed | 13 | 13 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Required Emergency Surgery | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants Who Received Study Drug: BAX326 : -Study Part 1: Pharmacokinetic (PK) Crossover with BAX326 and BeneFIX -Study Part 2: Open-label evaluation of prophylaxis and on-demand BAX326 only -Study Part 3: Open-label repeat of PK evaluation (repeat Study Part 1) with BAX326 only and same study participants as Study Part 1
Arm/Group | All Study Participants Who Received Study Drug
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 73
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 1
  Ukraine | 8
  Chile | 4
  Russian Federation | 12
  Colombia | 5
  United Kingdom | 2
  Czech Republic | 2
  Argentina | 2
  Brazil | 1
  Poland | 12
  Romania | 8
  Bulgaria | 10
  Japan | 5
  Sweden | 1

OUTCOME MEASURES:

1. Primary Outcome: Study Part 1- Area Under the Plasma Concentration Versus Time Curve From 0 to 72 Hours Per Dose
Description: Computed using the linear trapezoidal method. The concentration at 72 hours was interpolated from the two nearest sampling time points or extrapolated using the last quantifiable concentration and the terminal rate constant λz. λz was estimated from the slope of natural log-linear fitting to latter quantifiable concentrations, with largest adjusted R^2.
Time Frame: 72 hours
Population: Pharmacokinetic Per Protocol Analysis Set (PKPPAS) -Participants who participated in Study Parts 1-3 and completed Study Part 1 without any major protocol deviations
Measure: Median (Inter-Quartile Range); unit: (IU·hr/dL) / (IU/kg)
Arm/Group | BAX326 | BeneFIX
Number analyzed (Participants) | 25 | 25
(IU·hr/dL) / (IU/kg) | 14.30 [11.20 to 15.95] | 13.42 [11.08 to 15.10]
Statistical Analysis 1: Comparison: BAX326 vs BeneFIX; Test type: Non-Inferiority or Equivalence — Bioequivalence will be established if 90% C.I. of ratio is contained completely in the margins of equivalence of 0.8 to 1.25; Ratio of Geometric Means = 1.063, 90% CI 2-sided [1.03 to 1.09]

2. Secondary Outcome: Study Parts 1 and 3: Area Under the Plasma Concentration/Time Curve From Time 0 to Infinity Per Dose (AUC0-∞/ Dose)
Description: Defined as (AUC0-t + Ct)/ λz/ dose, where t is the time of last quantifiable concentration, Ct is the last quantifiable concentration. λz will be estimated from the slope of natural log-linear fitting to latter quantifiable concentrations, with largest adjusted R^2. The objective of Study Part 3 was to re-evaluate the Pharmacokinetic (PK) parameters for BAX 326 after a period of 6 months of treatment, in participants who accumulated at least 30 EDs to BAX 326, and to compare them with those determined in the same participants participating in Study Part 1.
Time Frame: 0-30 minutes before infusion up to 72 hours post-infusion
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: (IU·hr)/ dL/ (IU/kg)
Groups:
- Study Part 1: BAX326: PK infusion with BAX326 at 75 ± 5 IU/kg
- Study Part 1: BeneFIX: PK infusion with BeneFIX at 75 ± 5 IU/kg
- Study Part 3: BAX326: PK infusion with BAX326 at 75 ± 5 IU/kg Study Part 3 only evaluated BAX326 (ie BeneFIX was not evaluated in Study Part 3)
Arm/Group | Study Part 1: BAX326 | Study Part 1: BeneFIX | Study Part 3: BAX326
Number analyzed (Participants) | 25 | 25 | 23
(IU·hr)/ dL/ (IU/kg) | 16.07 [13.43 to 17.48] | 15.26 [13.71 to 17.05] | 17.38 [14.17 to 20.70]

3. Secondary Outcome: Study Parts 1 and 3: Mean Residence Time (MRT)
Description: Computed as Area under the moment curve 0-∞ (AUMC0-∞) / AUC0-∞- TI/2, where AUMC0-∞ will be determined in a similar manner as AUC0-∞ and TI represents infusion duration [hr] The objective of Study Part 3 was to re-evaluate the Pharmacokinetic (PK) parameters for BAX 326 after a period of 6 months of treatment, in participants who accumulated at least 30 EDs to BAX 326, and to compare them with those determined in the same participants participating in Study Part 1.
Time Frame: 0-30 minutes before infusion up to 72 hours post-infusion
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hour
Arm/Group | Study Part 1: BAX326 | Study Part 1: BeneFIX | Study Part 3: BAX326
Number analyzed (Participants) | 25 | 25 | 23
Hour | 28.93 [26.45 to 31.50] | 30.59 [28.13 to 34.84] | 29.04 [28.00 to 32.31]

4. Secondary Outcome: Study Parts 1 and 3: Clearance (CL)
Description: Computed as Dose/ AUC0-∞. The objective of Study Part 3 was to re-evaluate the Pharmacokinetic (PK) parameters for BAX 326 after a period of 6 months of treatment, in participants who accumulated at least 30 EDs to BAX 326, and to compare them with those determined in the same participants participating in Study Part 1.
Time Frame: 0-30 minutes before infusion up to 72 hours post-infusion
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: dL/(kg·hr)
Arm/Group | Study Part 1: BAX326 | Study Part 1: BeneFIX | Study Part 3: BAX326
Number analyzed (Participants) | 25 | 25 | 23
dL/(kg·hr) | 0.0622 [0.0572 to 0.0745] | 0.0655 [0.0587 to 0.0730] | 0.0576 [0.0483 to 0.0706]

5. Secondary Outcome: Study Parts 1 and 3: Incremental Recovery at Cmax (IR at Cmax)
Description: Defined as (Cmax - Cpre-infusion)/Dose, where maximum concentration (Cmax) will be determined as the highest concentration achieved within one hour after infusion. The objective of Study Part 3 was to re-evaluate the Pharmacokinetic (PK) parameters for BAX 326 after a period of 6 months of treatment, in participants who accumulated at least 30 EDs to BAX 326, and to compare them with those determined in the same participants participating in Study Part 1.
Time Frame: 0-30 minutes before infusion up to 1 hour post-infusion
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: (IU/dL) / (IU/kg)
Arm/Group | Study Part 1: BAX326 | Study Part 1: BeneFIX | Study Part 3: BAX326
Number analyzed (Participants) | 25 | 25 | 23
(IU/dL) / (IU/kg) | 0.88 [0.79 to 0.98] | 0.73 [0.66 to 0.87] | 0.93 [0.76 to 1.18]

6. Secondary Outcome: Incremental Recovery (IR) at 30 Minutes Over Time
Description: IR at 30 Minutes was measured at the following time points during the study: - Part 1 or Part 2, Exposure Day (ED) 1. (If participant was present for Study Part 1, then ED 1 from Part 1 was used. If Participant entered study in Study Part 2, then ED 1 from Part 2 was used.) - Part 2: Week 5 - Part 2: Week 13 - Part 2 or Part 3: Week 26 (Week 26 of study participation) - Study Completion or Termination Visit
Time Frame: 0-30 minutes before infusion and 30 minutes post-infusion
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: (IU/dL) / (IU/kg)
Groups:
- Part 1 or Part 2, ED 1: PK infusion with BAX326 at 75 ± 5 IU/kg
- Part 2: Week 5: PK infusion with BeneFIX at 75 ± 5 IU/kg
- Part 2: Week 13: PK infusion with BAX326 at 75 ± 5 IU/kg Study Part 3 only evaluated BAX326 (ie BeneFIX was not evaluated in Study Part 3)
Arm/Group | Part 1 or Part 2, ED 1 | Part 2: Week 5 | Part 2: Week 13 | Part 2 or Part 3: Week 26 | Study Completion or Termination Visit
Number analyzed (Participants) | 73 | 71 | 68 | 55 | 23
(IU/dL) / (IU/kg) | 0.78 [0.7 to 0.91] | 0.79 [0.68 to 0.96] | 0.83 [0.655 to 1.015] | 0.88 [0.75 to 1.04] | 0.89 [0.73 to 0.96]

7. Secondary Outcome: Change in Incremental Recovery (IR) at 30 Minutes Over Time
Description: The median changes in IR at 30 Minutes, calculated as the change in IR value from exposure day 1 (ED1).
Time Frame: 0-30 minutes before infusion and 30 minutes post-infusion
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: (IU/dL) / (IU/kg)
Groups:
- Part 2: Week 5: PK infusion with BAX326 at 75 ± 5 IU/kg
Arm/Group | Part 2: Week 5 | Part 2: Week 13 | Part 2 or Part 3: Week 26 | Study Completion or Termination Visit
Number analyzed (Participants) | 71 | 68 | 55 | 23
(IU/dL) / (IU/kg) | 0.03 [-0.09 to 0.11] | 0.075 [-0.07 to 0.17] | 0.06 [0.02 to 0.17] | 0.12 [0 to 0.21]

8. Secondary Outcome: Study Parts 1 and 3: Half Life (T 1/2)
Description: Elimination phase half-life will be determined as ln2/ λz. The objective of Study Part 3 was to re-evaluate the Pharmacokinetic (PK) parameters for BAX 326 after a period of 6 months of treatment, in participants who accumulated at least 30 EDs to BAX 326, and to compare them with those determined in the same participants participating in Study Part 1.
Time Frame: 0-30 minutes before infusion up to 72 hours post-infusion
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hour
Arm/Group | Study Part 1: BAX326 | Study Part 1: BeneFIX | Study Part 3: BAX326
Number analyzed (Participants) | 25 | 25 | 23
Hour | 24.58 [20.98 to 29.68] | 26.28 [22.51 to 29.46] | 24.59 [19.68 to 29.14]

9. Secondary Outcome: Study Parts 1 and 3: Volume of Distribution at Steady State (Vss)
Description: Vss computed as CL·MRT. The objective of Study Part 3 was to re-evaluate the Pharmacokinetic (PK) parameters for BAX 326 after a period of 6 months of treatment, in participants who accumulated at least 30 EDs to BAX 326, and to compare them with those determined in the same participants participating in Study Part 1.
Time Frame: 0-30 minutes before infusion up to 72 hours post-infusion
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: dL/kg
Arm/Group | Study Part 1: BAX326 | Study Part 1: BeneFIX | Study Part 3: BAX326
Number analyzed (Participants) | 25 | 25 | 23
dL/kg | 1.72 [1.56 to 2.30] | 1.98 [1.76 to 2.51] | 1.74 [1.49 to 2.05]

10. Secondary Outcome: Study Part 2: Annualized Bleed Rate (ABR) During Treatment With BAX326
Description: ABR during prophylaxis (twice-weekly) in Part 2 was calculated as (Number of bleeding episodes/observed treatment period in days) * 365.25. The treatment period on prophylaxis was defined as time between the first and the last prophylactic infusions and ABR on prophylaxis was calculated for participants who received a minimum of 3 months of prophylactic treatment with BAX326.
Time Frame: Study Part 2 = 26 weeks ± 1 week (Note: Study Part 1 = 2-4 weeks)
Population: Full Analysis Set - Prophylactic cohort
Measure: Median (Inter-Quartile Range); unit: Bleeds per year
Groups:
- BAX326 Prophylaxis: Prophylactic treatment of 50 IU/kg BAX326 twice weekly. The dose range is 40-60 IU/kg and may be increased up to 75 IU/kg, if required. Participants received a minimum of three months prophylactic treatment
Arm/Group | BAX326 Prophylaxis
Number analyzed (Participants) | 56
Bleeds per year
  Joint bleeding episode | 0.00 [0.0 to 4.5]
  Non-Joint bleeding episode | 0.00 [0.0 to 2.0]
  Spontaneous bleeding episode | 0.00 [0.0 to 2.0]
  Bleeding episode caused by injury | 0.00 [0.0 to 2.1]
  Unknown cause of bleeding episode | 0.00 [0.0 to 0.0]
  All bleeding episodes | 1.99 [0.0 to 6.5]

11. Secondary Outcome: Bleeding Episodes Treated With 1, 2 or ≥3 Infusions of BAX326 by Bleeding Site and Cause
Description: The number of bleeding episodes treated with 1, 2, or ≥3 infusions of BAX326 to achieve adequate hemostasis. Only infusions required until resolution of bleed were considered.
Time Frame: Study Part 2 = 26 weeks ± 1 week (Study Part 2 began at week 3-5)
Population: Full Analysis Set
Measure: Number; unit: Bleeding episodes
Units Other Than Participants: bleeding episodes
Arm/Group | Bleeding Site: Target Joint | Bleeding Site: Non-Target Joint | Bleeding Site: All Joint | Bleeding Site: Non-Joint | Bleeding Cause: Spontaneous | Bleeding Cause: Injury | Bleeding Cause: Unknown
Number analyzed (Participants) | 73 | 73 | 73 | 73 | 73 | 73 | 73
Number analyzed (bleeding episodes) | 107 | 90 | 197 | 52 | 130 | 90 | 29
Bleeding episodes
  1 infusion | 65 | 57 | 122 | 31 | 84 | 50 | 19
  2 infusions | 26 | 21 | 47 | 11 | 29 | 24 | 5
  3 or more infusions | 16 | 12 | 28 | 10 | 17 | 16 | 5

12. Secondary Outcome: Hemostatic Efficacy at Resolution of All Bleeding Episodes (BEs) Treated With BAX326 by Bleeding Site and Cause
Description: Rating Scale for Treatment of BEs (4-point ordinal scale): -Excellent: Full relief of pain and cessation of objective signs of bleeding (eg, swelling, tenderness, and decreased range of motion in the case of musculoskeletal hemorrhage) after a single infusion. No additional infusion required for the control of bleeding. Administration of further infusions to maintain hemostasis did not affect this scoring. -Good: Definite pain relief and/or improvement in signs of bleeding after a single infusion. Possibly requires more than 1 infusion for complete resolution. -Fair: Probable and/or slight relief of pain and slight improvement in signs of bleeding after single infusion. Required more than 1 infusion for complete resolution. -None: No improvement or condition worsens.
Time Frame: At bleed resolution throughout the study period of 22 months (Study Parts 1, 2, and 3)
Population: Full Analysis Set
Measure: Number; unit: Bleeding episodes
Units Other Than Participants: Bleeding episodes
Arm/Group | Bleeding Site: Target Joint | Bleeding Site: Non-Target Joint | Bleeding Site: All Joint | Bleeding Site: Non-Joint | Bleeding Cause: Spontaneous | Bleeding Cause: Injury | Bleeding Cause: Unknown
Number analyzed (Participants) | 73 | 73 | 73 | 73 | 73 | 73 | 73
Number analyzed (Bleeding episodes) | 107 | 90 | 197 | 52 | 130 | 90 | 29
Bleeding episodes
  Excellent | 53 | 32 | 85 | 17 | 51 | 40 | 11
  Good | 46 | 57 | 103 | 34 | 75 | 45 | 17
  Fair | 5 | 0 | 5 | 0 | 2 | 2 | 1
  None | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Reported | 3 | 1 | 4 | 1 | 2 | 3 | 0

13. Secondary Outcome: Total Weight-adjusted Dose Per Bleeding Episode (BEs) of All BEs Treated With BAX326 by Bleeding Site and Cause
Time Frame: Study Part 2 = 26 weeks ± 1 week (Note: Study Part 1 = 2-4 weeks)
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: IU/kg
Units Other Than Participants: Bleeding Episodes
Arm/Group | Bleeding Site: Target Joint | Bleeding Site: Non-Target Joint | Bleeding Site: All Joint | Bleeding Site: Non-Joint | Bleeding Cause: Spontaneous | Bleeding Cause: Injury | Bleeding Cause: Unknown
Number analyzed (Participants) | 73 | 73 | 73 | 73 | 73 | 73 | 73
Number analyzed (Bleeding Episodes) | 107 | 90 | 197 | 52 | 130 | 90 | 29
IU/kg | 56.5 [48 to 97] | 59.0 [46 to 97] | 56.5 [47 to 97] | 68.7 [50 to 130] | 52.3 [45 to 92] | 70.0 [48 to 116] | 56.5 [51 to 108]

14. Secondary Outcome: Consumption of BAX326 Per Event Per Participant
Description: Weight-adjusted consumption of BAX326 by event per participant, i.e., for prophylactic treatment and for treatment of bleeds until resolution of bleed.
Time Frame: Study Part 2 = 26 weeks ± 1 week (Note: Study Part 1 = 2-4 weeks)
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: IU/kg
Groups:
- Bleeding Treatment: Includes all participants who received any infusions for bleeding treatment in the Full Analysis Set. (ie includes all On-demand arm (N=14) and 33 participants from the prophylaxis arm who experienced a bleeding episode)
Arm/Group | Prophylactic Treatment | Bleeding Treatment
Number analyzed (Participants) | 59 | 47
IU/kg | 50.5 [46 to 52] | 87.1 [56 to 125]

15. Secondary Outcome: Consumption of BAX326 Per Participant: Median Number of Infusions Per Month
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week (Prophylaxis and On-Demand period), Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Infusions
Groups:
- Prophylaxis; On-Demand: Study Part 2 Only
Arm/Group | Prophylaxis | On-Demand
Number analyzed (Participants) | 59 | 14
Infusions | 6.7 [6 to 7] | 2.7 [2 to 4]

16. Secondary Outcome: Consumption of BAX326 Per Participant: Median Weight-adjusted Consumption Per Month
Time Frame: as for outcome 15
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: IU/kg
Arm/Group | Prophylaxis | On-Demand
Number analyzed (Participants) | 59 | 14
IU/kg | 347.8 [320 to 396] | 167.3 [102 to 234]

17. Secondary Outcome: Number of Participants Who Developed Inhibitory Antibodies to Factor IX (FIX)
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
participants | 0

18. Secondary Outcome: Occurrence of Total Binding Antibodies of Indeterminate Specificity (Within Assay Variability)
Description: Occurrence of total binding antibodies of indeterminate specificity (within assay variability) to FIX, antibodies to CHO proteins and rFurin is defined by a dilution of 2 or less increase as compared to levels at screening visit (e.g. negative to 1:20 or 1:40).
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
participants
  Binding Antibody to Factor IX (FIX) | 6
  Antibody to Chinese hamster ovary (CHO) Protein | 0
  Antibody to recombinant Furin (rFurin) | 9

19. Secondary Outcome: Occurrence of Treatment Related Total Binding Antibodies
Description: Occurrence of treatment related total binding antibodies to Factor IX (FIX), antibodies to Chinese hamster ovary (CHO) proteins, and recombinant furin (rFurin) is defined by more than 2-dilution increase as compared to levels at screening visit and confirmed specificity (e.g. negative to 1:80)
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
participants
  Binding Antibody to Factor IX (FIX) | 0
  Antibody to Chinese hamster ovary (CHO) Protein | 0
  Antibody to recombinant Furin (rFurin) | 0

20. Secondary Outcome: Number of Participants Who Experienced Severe Allergic Reactions (e.g. Anaphylaxis)
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
participants | 0

21. Secondary Outcome: Number of Participants Who Experienced Thrombotic Events
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
participants | 0

22. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Parameters: Clinical Chemistry
Description: Clinically significant changes in chemistry assessments for Alanine Aminotransferase, Albumin, Alkaline Phosphatase, Aspartate Aminotransferase, Bicarbonate, Bilirubin, Blood Urea Nitrogen, Chloride, Glucose, Potassium, Protein (Serum), Sodium. Clinically Significant (CS) defined as: -1. The abnormal value constitutes an adverse event (AE) and, -2. The abnormal value is a symptom of or related to a disease that is already recorded as an AE in Case Report Form (CRF).
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
participants | 0

23. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Parameters: Hematology
Description: Clinically significant changes in hematology assessments for Basophils, Basophils/Leukocytes, Eosinophils, Eosinophils/Leukocytes, Erythrocyte Mean Corpuscular Hemoglobin Concentration, Erythrocyte Mean Corpuscular Volume, Erythrocytes, Hematocrit, Hemoglobin, Leukocytes, Lymphocytes, Lymphocytes/Leukocytes, Monocytes, Monocytes/Leukocytes, Neutrophils, Neutrophils/Leukocytes, Platelets,
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
participants | 0

24. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Parameters: Vital Signs
Description: Clinically significant changes in vital signs assessments for pulse rate, systolic/diastolic blood pressure, respiratory rate, body temperature
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
participants | 0

25. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Parameters: Thrombogenic Markers
Description: Clinically significant changes in thrombogenic markers assessments for thrombin-antithrombin (TAT), prothrombin fragment 1.2, and D-dimer as evaluated by an independent Data Monitoring Committee (DMC)
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
participants | 0

26. Secondary Outcome: Number of Adverse Events (AEs) After BAX326 Treatment
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, and Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Number; unit: adverse events
Groups:
- AEs - Related: Probable, possible, or unknown causality assessment of an AE will be counted as "related".
Arm/Group | AEs - Not Related | AEs - Related
Number analyzed (Participants) | 73 | 73
adverse events
  Serious- Mild | 1 | 0
  Serious- Moderate | 1 | 0
  Serious- Severe | 3 | 0
  Serious- Unknown | 0 | 0
  Non-Serious- Mild | 63 | 2
  Non-Serious- Moderate | 17 | 0
  Non-Serious- Severe | 1 | 0
  Non-Serious- Unknown | 1 | 1

27. Secondary Outcome: Number of Participants With Adverse Events (AEs) After BAX326 Treatment
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, and Study Part 3 = 1 week (Total = 29-31 weeks)
Measure: Number; unit: participants
Groups:
- Participants With AEs - Related: Probable, possible, or unknown causality assessment of an AE will be counted as "related".
Arm/Group | Participants With AEs - Not Related | Participants With AEs - Related
Number analyzed (Participants) | 73 | 73
participants
  Serious- Mild | 1 | 0
  Serious- Moderate | 1 | 0
  Serious- Severe | 2 | 0
  Serious- Unknown | 0 | 0
  Non-Serious- Mild | 33 | 1
  Non-Serious- Moderate | 9 | 0
  Non-Serious- Severe | 1 | 0
  Non-Serious- Unknown | 1 | 1

28. Secondary Outcome: EuroQoL (Quality of Life)-5 Dimensions (EQ-5D) Total Index Scores
Description: EQ-5D is a participant answered questionnaire scoring 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D total score ranges from 0 (worst health state) to 1 (perfect health state) and 1 reflects the best outcome.
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline): Prophylactic treatment of 50 IU/kg BAX326 twice weekly. The dose range is 40-60 IU/kg and may be increased up to 75 IU/kg, if required.
- On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline): On-Demand Dosing and Frequency (Guidance): • Early hemarthrosis, muscle bleed, oral bleed= FIX level required(%) 20-40 IU/dL. Repeat every 24 hours. Duration: at least 1 day, until bleeding episode as indicated by pain is resolved or healing is achieved • More extensive hemarthrosis, muscle bleed, hematoma= FIX level required(%) 30-60 IU/dL. Repeat infusion every 24 hours for 3-4 days or more until pain and acute disability are resolved • Life threatening hemorrhages= FIX level required(%) 60-100 IU/dL. Repeat infusion every 8-24 hours until threat resolves Required dose calculated using IR determined of first 16 participants who completed Part 1 according to: Body weight (kg) x desired FIX rise (%) (IU/dL) x {reciprocal of observed recovery} Given an anticipated recovery of 0.8 [IU/dl]/[IU/kg], required units calculated by: Body weight (kg) x desired FIX rise (%or (IU/dL) x 1.3 IU/kg Amount administered & frequency should be oriented to individual clinical effectiveness
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 56 | 55 | 55 | 14 | 14 | 14
Score on a scale | 0.75 (0.16) [0.7 to 0.8] | 0.75 (0.16) [0.7 to 0.8] | 0.01 (0.18) [-0.1 to 0.1] | 0.72 (0.14) | 0.73 (0.09) | 0.00 (0.13)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.7790, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) vs On-Demand: End of Study; Test type: Superiority or Other; p = 0.8999, Paired t-test

29. Secondary Outcome: EuroQoL (Quality of Life)-5 Dimensions Visual Analogue Scale (EQ-5D VAS) Scores
Description: Participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better quality of life.
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 56 | 54 | 54 | 14 | 14 | 14
Score on a scale | 58.75 (24.89) [50.0 to 75.0] | 68.22 (22.78) [60.0 to 85.0] | 9.98 (25.41) [-2.0 to 20.0] | 56.64 (25.97) | 62.07 (19.00) | 5.43 (24.02)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.0056, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) vs On-Demand: End of Study; Test type: Superiority or Other; p = 0.4130, Paired t-test

30. Secondary Outcome: General Pain Assessment Through a Visual Analog Scale (VAS)
Description: Participant rated assessment of health-related quality of life. The VAS Pain Scale rates current health state on a scale from 0 (no pain) to 100 (worst imaginable pain). For the pain scale, a higher score indicates worse pain.
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 55 | 55 | 54 | 14 | 14 | 14
Score on a scale | 32.67 (26.62) | 33.09 (25.90) | 0.35 (21.77) | 47.57 (30.82) | 39.93 (22.57) | -7.64 (33.58)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.9059, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) vs On-Demand: End of Study; Test type: Superiority or Other; p = 0.4098, Paired t-test

31. Secondary Outcome: Short Form (36) Health Survey (SF-36): HRQoL 'Physical Component Score' (PCS)
Description: The PCS is a summary scale of the dimensions physical functioning, role physical, bodily pain, and general health. The component score is normalized to a standard population. Scores range from 0 to 100 with higher scores representing better health. There is no total overall score; scoring is done for both subscores and summary scores.
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 54 | 52 | 52 | 13 | 13 | 13
Score on a scale | 39.08 (9.39) | 41.35 (8.73) | 2.60 (7.72) | 37.38 (7.20) | 38.92 (8.53) | 1.54 (5.11)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.0189, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) vs On-Demand: End of Study; Test type: Superiority or Other; p = 0.2974, Paired t-test

32. Secondary Outcome: SF-36: HRQoL 'Mental Health' (MH)
Description: Quality of life survey response as measured using the SF-36 questionnaire. Scores range from 0 to 100 with higher scores representing better health. There is no total overall score; scoring is done for both subscores and summary scores. The raw data from the SF-36 items were transformed to norm based scores for each of the 8 HRQoL/SF-36 health domain scores.
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 54 | 52 | 52 | 13 | 13 | 13
Score on a scale | 47.53 (9.46) | 49.67 (9.30) | 2.01 (11.17) | 47.24 (8.80) | 45.03 (9.96) | -2.21 (8.28)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.2009, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) vs On-Demand: End of Study; Test type: Superiority or Other; p = 0.3552, Paired t-test

33. Secondary Outcome: SF-36: HRQoL Physical Functioning' (PF)
Description: as for outcome 32
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 54 | 53 | 53 | 13 | 13 | 13
Score on a scale | 40.20 (10.57) | 40.75 (10.14) | 0.68 (7.48) | 40.04 (10.57) | 39.87 (10.55) | -0.16 (5.86)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.5143, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) vs On-Demand: End of Study; Test type: Superiority or Other; p = 0.9223, Paired t-test

34. Secondary Outcome: SF-36: HRQoL Role-Physical (RP)
Description: as for outcome 32
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 54 | 53 | 53 | 13 | 13 | 13
Score on a scale | 40.39 (10.70) | 43.82 (8.67) | 3.47 (10.15) | 39.15 (8.13) | 37.45 (10.12) | -1.70 (5.86)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.0162, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) vs On-Demand: End of Study; Test type: Superiority or Other; p = 0.3176, Paired t-test

35. Secondary Outcome: SF-36: HRQoL Role-Emotional
Description: as for outcome 32
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 54 | 53 | 53 | 13 | 13 | 13
Score on a scale | 44.22 (11.45) | 44.80 (10.15) | 0.37 (11.74) | 40.93 (9.10) | 39.43 (11.57) | -1.50 (8.91)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.8210, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) vs On-Demand: End of Study; Test type: Superiority or Other; p = 0.5565, Paired t-test

36. Secondary Outcome: SF-36: HRQoL Bodily Pain
Description: as for outcome 32
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 54 | 53 | 53 | 13 | 13 | 13
Score on a scale | 42.09 (10.21) | 45.72 (8.68) | 3.45 (9.95) | 36.89 (7.84) | 39.33 (8.91) | 2.44 (10.18)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.0146, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) vs On-Demand: End of Study; Test type: Superiority or Other; p = 0.4048, Paired t-test

37. Secondary Outcome: SF-36: HRQoL Mental Health
Description: as for outcome 32
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 54 | 52 | 52 | 13 | 13 | 13
Score on a scale | 45.52 (8.78) | 47.95 (8.84) | 2.44 (11.29) | 45.46 (10.57) | 42.64 (10.63) | -2.82 (8.53)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.1258, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) vs On-Demand: End of Study; Test type: Superiority or Other; p = 0.2567, Paired t-test

38. Secondary Outcome: SF-36: HRQoL Vitality
Description: as for outcome 32
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 54 | 52 | 52 | 13 | 13 | 13
Score on a scale | 50.07 (8.47) | 52.75 (8.88) | 2.46 (10.75) | 50.17 (5.63) | 50.89 (6.81) | 0.72 (5.43)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.1048, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) vs On-Demand: End of Study; Test type: Superiority or Other; p = 0.6410, Paired t-test

39. Secondary Outcome: SF-36: HRQoL Social Functioning
Description: as for outcome 32
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Prophylaxis: Part 1 or Part 2, Exposure Day (ED) 1 (Baseline): Prophylactic treatment of 50 IU/kg BAX326 twice weekly. The dose range is 40-60 IU/kg and may be increased up to 75 IU/kg, if required.
- On-Demand: Part 1 or Part 2, Exposure Day (ED) 1 (Baseline): On-Demand Dosing and Frequency (Guidance): • Early hemarthrosis, muscle bleed, oral bleed= FIX level required(%) 20-40 IU/dL. Repeat every 24 hours. Duration: at least 1 day, until bleeding episode as indicated by pain is resolved or healing is achieved • More extensive hemarthrosis, muscle bleed, hematoma= FIX level required(%) 30-60 IU/dL. Repeat infusion every 24 hours for 3-4 days or more until pain and acute disability are resolved • Life threatening hemorrhages= FIX level required(%) 60-100 IU/dL. Repeat infusion every 8-24 hours until threat resolves Required dose calculated using IR determined of first 16 participants who completed Part 1 according to: Body weight (kg) x desired FIX rise (%) (IU/dL) x {reciprocal of observed recovery} Given an anticipated recovery of 0.8 [IU/dl]/[IU/kg], required units calculated by: Body weight (kg) x desired FIX rise (%or (IU/dL) x 1.3 IU/kg Amount administered & frequency should be oriented to individual clinical effectiveness
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day (ED) 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day (ED) 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 54 | 53 | 53 | 13 | 13 | 13
Score on a scale | 41.80 (10.54) | 44.60 (8.94) | 2.78 (10.78) | 43.42 (9.61) | 42.17 (9.80) | -1.26 (6.36)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day (ED) 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.0663, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: Part 1 or Part 2, Exposure Day (ED) 1 (Baseline) vs On-Demand: End of Study; Test type: Superiority or Other; p = 0.4890, Paired t-test

40. Secondary Outcome: SF-36: HRQoL General Health
Description: as for outcome 32
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 54 | 53 | 53 | 13 | 13 | 13
Score on a scale | 37.84 (8.38) | 39.98 (9.03) | 2.20 (8.22) | 37.09 (10.47) | 39.07 (8.88) | 1.98 (7.94)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.0562, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: End of Study; Test type: Superiority or Other; p = 0.3864, Paired t-test

41. Secondary Outcome: Pediatric Quality of Life Questionnaire (PedsQL) Physical Health Summary Score (Ages 12-16)
Description: The Peds-QL is a generic Health-Related Quality of Life (HR QoL) instrument designed specifically for a pediatric population. It captures the following domains: general health/activities, feelings/emotional, social functioning, school functioning. For this study, the Peds-QL for 12 to 16-year-old subjects was used. Higher scores indicate better quality of life (QOL) for all domains of the Peds-QL. This modular instrument uses a 5-point scale: from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. 4 dimensions (physical, emotional, social, & school functioning) are scored.
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 2 | 2 | 2 | 1 | 1 | 1
Score on a scale | 65.63 (13.26) | 54.69 (6.63) | -10.94 (19.89) | 65.63 (NA) — Sample size = 1, therefore not possible to calculate a standard deviation. | 65.63 (NA) — Sample size = 1, therefore not possible to calculate a standard deviation. | 0.00 (NA) — Sample size = 1, therefore not possible to calculate a standard deviation.
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.5792, Paired t-test

42. Secondary Outcome: Pediatric Quality of Life Questionnaire (PedsQL) Psychosocial Health Summary Score (Ages 12-16)
Description: as for outcome 41
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 2 | 2 | 2 | 1 | 1 | 1
Score on a scale | 63.33 (11.79) | 55.83 (3.54) | -7.50 (8.25) | 88.33 (NA) — Sample size = 1, therefore not possible to calculate a standard deviation. | 86.67 (NA) — Sample size = 1, therefore not possible to calculate a standard deviation. | -1.67 (NA) — Sample size = 1, therefore not possible to calculate a standard deviation.
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.4208, Paired t-test

43. Secondary Outcome: Pediatric Quality of Life Questionnaire (PedsQL) Total Score (Ages 12-16)
Description: as for outcome 41
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 2 | 2 | 2 | 1 | 1 | 1
Score on a scale | 64.13 (12.30) | 55.43 (0.00) | -8.70 (12.30) | 80.43 (NA) — Sample size = 1, therefore not possible to calculate a standard deviation. | 79.35 (NA) — Sample size = 1, therefore not possible to calculate a standard deviation. | -1.09 (NA) — Sample size = 1, therefore not possible to calculate a standard deviation.
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.5000, Paired t-test

44. Secondary Outcome: Health-Related Quality of Life (HRQoL) Disease-specific: Haem-A-QoL
Description: The Haem-A-QOL instrument has been developed and used in hemophilia A patients. As a hemophilia-specific instrument, this measure assesses very specific aspects of dealing with hemophilia. The areas covered by this instrument are: physical health, sports/leisure, school/work, dealing with hemophilia, and outlook for the future. For the Haem-A-QOL, higher scores indicate a worse quality of life. Scores on a scale range between 0 and 100.
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) | Prophylaxis: End of Study | Prophylaxis: Change From Baseline | On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) | On-Demand: End of Study | On-Demand: Change From Baseline
Number analyzed (Participants) | 51 | 50 | 48 | 13 | 13 | 13
Score on a scale | 40.68 (15.33) | 37.85 (16.57) | -3.52 (12.81) | 41.65 (15.19) | 41.37 (16.64) | -0.28 (12.18)
Statistical Analysis 1: Comparison: Prophylaxis: Part 1 or Part 2, Exposure Day 1 (Baseline) vs Prophylaxis: End of Study; Test type: Superiority or Other; p = 0.0633, Paired t-test
Statistical Analysis 2: Comparison: On-Demand: Part 1 or Part 2, Exposure Day 1 (Baseline) vs On-Demand: End of Study; Test type: Superiority or Other; p = 0.9363, Paired t-test

45. Secondary Outcome: Health-Related Quality of Life (HRQoL) Disease-specific: Haemo-QoL - Participants On-Demand (Ages 12-16)
Description: The Haemo-QoL is a quality of life (QoL) assessment instrument for children and adolescents with haemophilia. As a hemophilia-specific instrument, this measure assesses very specific aspects of dealing with hemophilia. For the Haemo-QoL, higher scores indicate a worse quality of life. Scores on a scale range between 0 and 100.
Time Frame: Baseline at either Study Part 1, or Study Part 2, and End of Study (study weeks 29-31)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part 1 or Part 2, Exposure Day 1 (Baseline) | End of Study | Change From Baseline
Number analyzed (Participants) | 1 | 1 | 1
Score on a scale | 40.00 (NA) — Sample size = 1, therefore not possible to calculate a standard deviation. | 40.00 (NA) — Sample size = 1, therefore not possible to calculate a standard deviation. | 0.00 (NA) — Sample size = 1, therefore not possible to calculate a standard deviation.

46. Secondary Outcome: Health Resource Use - Number of Hospitalizations
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Median (Full Range); unit: Hospitalizations
Groups:
- Prophylaxis: Prophylactic treatment of 50 IU/kg BAX326 twice weekly. The dose range is 40-60 IU/kg and may be increased up to 75 IU/kg, if required.
- On-Demand: On-Demand Dosing and Frequency (Guidance): • Early hemarthrosis, muscle bleed, oral bleed= FIX level required(%) 20-40 IU/dL. Repeat every 24 hours. Duration: at least 1 day, until bleeding episode as indicated by pain is resolved or healing is achieved • More extensive hemarthrosis, muscle bleed, hematoma= FIX level required(%) 30-60 IU/dL. Repeat infusion every 24 hours for 3-4 days or more until pain and acute disability are resolved • Life threatening hemorrhages= FIX level required(%) 60-100 IU/dL. Repeat infusion every 8-24 hours until threat resolves Required dose calculated using IR determined of first 16 participants who completed Part 1 according to: Body weight (kg) x desired FIX rise (%) (IU/dL) x {reciprocal of observed recovery} Given an anticipated recovery of 0.8 [IU/dl]/[IU/kg], required units calculated by: Body weight (kg) x desired FIX rise (%or (IU/dL) x 1.3 IU/kg Amount administered & frequency should be oriented to individual clinical effectiveness
Arm/Group | Prophylaxis | On-Demand
Number analyzed (Participants) | 57 | 14
Hospitalizations
  Part 1 - Pharmacokinetics (N= 28, NA) | 0.0 [0 to 0] | NA [NA to NA] — There were no participants from the On-Demand arm in Study Part 1
  Part 2: Exposure Day 1 (N= 31, 14) | 0.0 [0 to 0] | 0.0 [0 to 0]
  Part 2: Week 5 (N= 57, 14) | 0.0 [0 to 1] | 0.0 [0 to 0]
  Part 2: Week 13 (N= 56, 12) | 0.0 [0 to 1] | 0.0 [0 to 0]
  Part 2: Week 26 (N= 30, NA) | 0.0 [0 to 0] | NA [NA to NA] — There were no participants from the On-Demand arm in Study Part 2 at Week 26
  Part 3 (N= 25, NA) | 0.0 [0 to 3] | NA [NA to NA] — There were no participants from the On-Demand arm in Study Part 3
  Completion/Termination (N= 20, 9) | 0.0 [0 to 1] | 0.0 [0 to 0]
  Unscheduled Study Visit (N= 1, NA) | 0.0 [0 to 0] | NA [NA to NA] — There were no participants from the On-Demand arm with an unscheduled Study Visit

47. Secondary Outcome: Health Resource Use - Total Days of Hospital Stay
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Median (Full Range); unit: Days
Arm/Group | Prophylaxis
Number analyzed (Participants) | 4
Days
  Part 2: Week 5 (N= 1) | 46.0 [46 to 46]
  Part 2: Week 13 (N= 1) | 23.0 [23 to 23]
  Part 3 (N= 3) | 2.0 [1 to 16]
  Completion/Termination (N= 2) | 5.5 [2 to 9]

48. Secondary Outcome: Health Resource Use - Emergency Room Visits
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Median (Full Range); unit: Visits
Arm/Group | Prophylaxis | On-Demand
Number analyzed (Participants) | 57 | 14
Visits
  Part 1 - Pharmacokinetics (N= 28, NA) | 0.0 [0 to 0] | NA [NA to NA] — There were no participants from the On-Demand arm in Study Part 1
  Part 2: Exposure Day 1 (N= 31, 14) | 0.0 [0 to 10] | 0.0 [0 to 0]
  Part 2: Week 5 (N= 57, 14) | 0.0 [0 to 1] | 0.0 [0 to 0]
  Part 2: Week 13 (N= 56, 12) | 0.0 [0 to 1] | 0.0 [0 to 0]
  Part 2: Week 26 (N= 30, NA) | 0.0 [0 to 0] | NA [NA to NA] — There were no participants from the On-Demand arm in Study Part 2 at Week 26
  Part 3 (N= 25, NA) | 0.0 [0 to 0] | NA [NA to NA] — There were no participants from the On-Demand arm in Study Part 3
  Completion/Termination (N= 20, 9) | 0.0 [0 to 1] | 0.0 [0 to 0]
  Unscheduled Study Visit (N= 1, NA) | 0.0 [0 to 0] | NA [NA to NA] — There were no participants from the On-Demand arm with an unscheduled Study Visit

49. Secondary Outcome: Health Resource Use - Unscheduled Doctor's Office Visits
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Median (Full Range); unit: Visits
Arm/Group | Prophylaxis | On-Demand
Number analyzed (Participants) | 57 | 14
Visits
  Part 1 - Pharmacokinetics (N= 28, NA) | 0.0 [0 to 1] | NA [NA to NA] — There were no participants from the On-Demand arm in Study Part 1
  Part 2: Exposure Day 1 (N= 31, 14) | 0.0 [0 to 0] | 0.0 [0 to 0]
  Part 2: Week 5 (N= 57, 14) | 0.0 [0 to 3] | 0.0 [0 to 0]
  Part 2: Week 13 (N= 56, 12) | 0.0 [0 to 2] | 0.0 [0 to 0]
  Part 2: Week 26 (N= 30, NA) | 0.0 [0 to 1] | NA [NA to NA] — There were no participants from the On-Demand arm in Study Part 2 at Week 26
  Part 3 (N= 25, NA) | 0.0 [0 to 1] | NA [NA to NA] — There were no participants from the On-Demand arm in Study Part 3
  Completion/Termination (N= 20, 9) | 0.0 [0 to 2] | 0.0 [0 to 1]
  Unscheduled Study Visit (N= 1, NA) | 1.0 [1 to 1] | NA [NA to NA] — There were no participants from the On-Demand arm with an unscheduled Study Visit

50. Secondary Outcome: Health Resource Use - Days Lost From Work or School
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Population: Full Analysis Set
Measure: Median (Full Range); unit: Days
Arm/Group | Prophylaxis | On-Demand
Number analyzed (Participants) | 57 | 14
Days
  Part 1 - Pharmacokinetics (N= 28, NA) | 0.0 [0 to 10] | NA [NA to NA] — There were no participants from the On-Demand arm in Study Part 1
  Part 2: Exposure Day 1 (N= 31, 14) | 0.0 [0 to 2] | 0.0 [0 to 0]
  Part 2: Week 5 (N= 57, 14) | 0.0 [0 to 8] | 0.0 [0 to 4]
  Part 2: Week 13 (N= 56, 12) | 0.0 [0 to 7] | 0.0 [0 to 0]
  Part 2: Week 26 (N= 30, NA) | 0.0 [0 to 5] | NA [NA to NA] — There were no participants from the On-Demand arm in Study Part 2 at Week 26
  Part 3 (N= 25, NA) | 0.0 [0 to 1] | NA [NA to NA] — There were no participants from the On-Demand arm in Study Part 3
  Completion/Termination (N= 20, 9) | 0.0 [0 to 24] | 0.0 [0 to 0]
  Unscheduled Study Visit (N= 1, NA) | 0.0 [0 to 0] | NA [NA to NA] — There were no participants from the On-Demand arm with an unscheduled Study Visit

ADVERSE EVENTS:
Time Frame: Study Part 1 = 2-4 weeks, Study Part 2 = 26 weeks ± 1 week, Study Part 3 = 1 week (Total = 29-31 weeks)
Groups:
- BAX326: BAX326: -Study Part 1: Pharmacokinetic (PK) Crossover with BAX326 and BeneFIX •Study Part 2: Open-label evaluation of prophylaxis and on-demand BAX326 only •Study Part 3: Open-label repeat of PK evaluation (repeat Study Part 1) with BAX326 only and same study participants as Study Part 1
Arm/Group | BAX326
Serious Adverse Events (participants affected / at risk) | 4/73
Other Adverse Events (participants affected / at risk) | 15/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAX326 (N=73)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Hepatitis B Core Antibody Positive (Investigations) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAX326 (N=73)
Nasopharyngitis (Infections and infestations) | 6 (8)
Immunology Test Abnormal (Investigations) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements may vary with individual PIs, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or up to 3 years after study completion. Baxter requires a review of results communications (eg for confidential information) ≥60 days prior to submission/communication. Baxter may request additional delay of ≤180 days(e.g., for intellectual property protection). Prior authorization may be required.